CLINICAL TRIAL: NCT00864643
Title: A Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of TAK-475 (100 mg) Vs Placebo When Coadministered With Atorvastatin (10 or 20 mg) in Subjects With Primary Hypercholesterolemia
Brief Title: Efficacy and Safety of Lapaquistat Acetate Coadministered With Atorvastatin in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-475-011; U1111-1122-7848 (Registry Identifier: WHO)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 100 mg QD + Atorvastatin QD (Experimental)
  Interventions: Drug: Lapaquistat acetate and atorvastatin
- Atorvastatin QD (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate and atorvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and atorvastatin 10 mg or 20 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: Lapaquistat acetate; Lipitor; TAK-475
  Arms: Lapaquistat Acetate 100 mg QD + Atorvastatin QD
Drug: Atorvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and atorvastatin 10 mg or 20 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: Lipitor; TAK-475
  Arms: Atorvastatin QD

SUMMARY:
The purpose of this study is to determine the efficacy of lapaquistat acetate, once daily (QD), coadministered with a statin to lower lipid levels in Subjects with Hypercholesterolemia.

DETAILED DESCRIPTION:
Elevated plasma cholesterol (hypercholesterolemia) and various other plasma lipid imbalances (dyslipidemias) are major risk factors for coronary heart disease. Normally, the balance among cholesterol synthesis, dietary intake, and degradation is adequate to maintain healthy cholesterol plasma levels. However, in patients with hypercholesterolemia, elevation in low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls. Consequently, it has been established that lowering the low-density lipoprotein cholesterol plasma concentration effectively reduces cardiovascular morbidity and mortality. As a result of this finding, the National Cholesterol Education Program Adult Treatment Panel III identifies control of low-density lipoprotein cholesterol as essential in the prevention and management of coronary heart disease. Additional lipid risk factors designated by Adult Treatment Panel III include elevated triglycerides, elevated non-high density lipoprotein cholesterol, and low levels of high-density lipoprotein cholesterol. Lipoproteins rich in triglycerides, such as very low-density lipoprotein cholesterol, appear to contribute to atherosclerosis, whereas the apparent protective effect of high-density lipoprotein cholesterol may be limited at low density lipoprotein concentrations.

TAK-475 (lapaquistat acetate) is a squalene synthase inhibitor currently under development at Takeda for the treatment of dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Prior to Screening, participant is not taking any lipid lowering agents and has an low-density lipoprotein cholesterol greater than 145 mg/dL and triglycerides less than 400 mg/dL, or is taking atorvastatin (10 mg or 20 mg) and has an low-density lipoprotein cholesterol greater than 100 mg/dL and triglycerides less than 400 mg/dL.
* Prior to Randomization, participant has taken at least 80% of open-label atorvastatin (10 mg or 20 mg) doses during Run-in, and has a mean low-density lipoprotein cholesterol greater than or equal to 100 mg/dL for 2 consecutive samples within 15% of each other.

Exclusion Criteria:

* Has been in remission for at least 5 years prior to the first dose of study drug. This criterion did not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.
* Has an alanine aminotransferase and aspartate aminotransferase level of greater than 1.5x the upper limit of normal, creatine phosphokinase greater than 3 times the upper limit of normal, active liver disease, jaundice, or serum creatinine greater than 2.0 mg/dL (men) or 1.8 mg/dL (women) at Screening.
* Has diabetes or a history of liver disease or had a positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history and/or subject's verbal report.
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain and/or discontinuation of statin due to myalgia.
* Has a positive human immunodeficiency virus status or had been taking retroviral medications, as determined by medical history and/or subject's verbal report.
* Has a body mass index of less than 15 or greater than 35 (weight/height2).
* Has a history of drug abuse or a history of alcohol abuse.
* Is currently participating in another investigational study or has participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* Has any other serious disease or condition at Screening or at Randomization that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.
* Has a known hypersensitivity or history of adverse reaction to lapaquistat acetate, atorvastatin or other statins, or multiple intolerances or allergies to other medications.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Lipid-lowering agents (including cholesterol absorption inhibitors, ethylicosapentate, plant sterols, niacin, and fibrates).
  * Any statin, other than atorvastatin

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2004-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in Low Density Lipoprotein Cholesterol | Week 6

SECONDARY OUTCOMES:
Percent change from Baseline in Total Cholesterol | Week 6
Percent change from Baseline in High-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in Triglycerides | Week 6
Percent change from Baseline in Apolipoprotein B | Week 6
Percent change from Baseline in Apolipoprotein A1 | Week 6
Percent change from Baseline in Very-Low Density Lipoprotein Cholesterol | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Science Strategy, Study Director — Takeda

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985